CLINICAL TRIAL: NCT05401994
Title: Screw Retained Arch Bar Versus Conventional Erich's Arch Bar in Maxillomandibular Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A03080921
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-05

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional Erich's arch bar (Active Comparator): • Patients will receive conventional Erich's arch bar
  Interventions: Procedure: conventional Erich's Arch Bar
- Screw Retained Arch Bar (Experimental): patients will receive modified screw retained arch bar.
  Interventions: Procedure: screw retained arch bar

INTERVENTIONS:
Procedure: screw retained arch bar — maxillomandibular fixation with bone screwed arch bar
  Arms: Screw Retained Arch Bar
Procedure: conventional Erich's Arch Bar — maxillomandibular fixation with conventional arch bar fixed to the teeth
  Arms: conventional Erich's arch bar

SUMMARY:
A randomized prospective clinical study to compare screw Retained Arch Bar and Conventional Erich's Arch Bar in Maxillomandibular Fixation

DETAILED DESCRIPTION:
2) Patients with non-pathological favorable or non-favorable fracture of mandible or maxilla that can be treated by MMF when acceptable occlusion can be obtained via bimanual reduction will be divided randomly into two equal groups: Group I: 10 patients will receive conventional Erich's arch bar. Group II: 10 patients will receive modified screw retained arch bar.

ELIGIBILITY:
Inclusion Criteria:

1. The patients age ranges from 18 to 50 years.
2. Patients with non-pathological favorable or non-favorable fracture of mandible or maxilla that can be treated by MMF when acceptable occlusion can be obtained via bimanual reduction.
3. Patients medically free from any systemic disease that absolutely contraindicate the surgical procedures.

Exclusion Criteria:

* 1) Edentulous ridge fracture. 2) Patients having primary and mixed dentition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
duration of surgical procedure in minutes | intraoperative
  Duration between the starting of fixation and complete fixation of fracture
maxillomandibular fixation stability in nominal scale(stable-unstable) | immediately postoperative
  stability after fixation
maxillomandibular fixation stability in nominal scale(stable-unstable) | 4-6 weeks
  stability after fixation
oral hygiene measuring with Oral Hygiene Index-Simplified (OHI-S) | immediately postoperative
  the OHI-S values range from 0 to 6.OHI-S score is good between 0 and 1.2, medium between 1.3 and 3, and poor between 3.1 and 6.
oral hygiene measuring with Oral Hygiene Index-Simplified (OHI-S) | 4-6 weeks
  the OHI-S values range from 0 to 6.OHI-S score is good between 0 and 1.2, medium between 1.3 and 3, and poor between 3.1 and 6.

SECONDARY OUTCOMES:
number of iatrogenic injuries | intraoperative
  iatrogenic injuries to teeth and gingiva
number of needle and wire stick injuries | intraoperative
  injuries to the surgeon and the assistants.
pain assessment using numeric rating scale (NRS) | immediately postoperative
  participants rated their pain on a scale from 0 to 10. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No